CLINICAL TRIAL: NCT00334295
Title: An Open, Non-randomised Multicentre Phase II Study to Assess the Efficacy and Tolerability of a 250 mg Monthly Dose of i.m. Applied Fulvestrant for the Treatment of Recurrent or Metastatic Endometrial Carcinoma.
Brief Title: Fulvestrant for the Treatment of Recurrent or Metastatic Endometrial Carcinoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9238GR/0002
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-06

CONDITIONS: Endometrial Carcinoma
Keywords: Recurrent or metastatic endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — A monthly intramuscular application of 250 mg Fulvestrant as a 1st line endocrine therapy in patients with recurrent or metastatic endometrial carcinoma.

SUMMARY:
The purpose of this study is to determine the efficacy of a monthly administration of Fulvestrant in patients with recurrent or metastatic endometrial carcinoma by assessment of the clinical tumour response after 3 injections.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, recurrent or metastatic endometrial carcinoma
* Postmenopausal
* Hormonreceptor positive

Exclusion Criteria:

* Pre-treatment with Fulvestrant
* Previous endocrine therapy of the endometrial carcinoma
* Previous malignancy less than 3 years ago other than in situ carcinoma of the cervix, basal cell carcinoma or squamous carcinoma of the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, MD, Study Director — AstraZeneca
Locations (9):
- Germany (9):
  - Research Site, Erlangen
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Jena
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Neunkirchen
  - Research Site, Rostock

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fulvestrant
Started | 35
Completed | 30
Not Completed | 5
Not completed — Patients received fewer than 3 injection | 5

BASELINE CHARACTERISTICS:
Arm/Group | Fulvestrant
Number analyzed (Participants) | 35
Age, Customized [Median (Full Range); unit: years] — post-menopausal
  years | 69.5 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Determination (for ITT (Intet-to-Treat Set): Efficacy of a Monthly Administration of Fulvestrant in Patients With Recurrent or Metastatic Endometrial Carcinoma by Assessment of the Clinical Tumour Response After 3 Injections of Fulvestrant
Description: Number of patients with Complete Remission (CR) and Partial Response (PR), as determined by an independent expert panel according to the WHO response criteria.
Time Frame: up to 1 year
Measure: Number; unit: participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 26
participants | 5

2. Secondary Outcome: Time to Progression of Disease (TTP-Time To Progression, for ITT Set)
Description: median TTP
Time Frame: ICF (Informed Consent Form completed) to the date of objective progression or death (by any cause in the absence of progression)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant
Number analyzed (Participants) | 26
months | 3.1 [2.6 to 6.5]

3. Secondary Outcome: Determination (for ITT Set): Median Survival
Description: median overall survival (OS)
Time Frame: ICF to the date of death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant
Number analyzed (Participants) | 26
months | 16.7 [8.6 to 44.4]

4. Secondary Outcome: Determination (All Subjects Treated (AST) Set): Safety and Toxicity by Assessment of the Frequency of Grade I-IV Haematological and Non-haematological Toxicities
Description: number of adverse events
Time Frame: ICF to Last Patient Out (LPO)
Measure: Number; unit: adverse events
Arm/Group | Fulvestrant
Number analyzed (Participants) | 35
adverse events | 169

5. Secondary Outcome: Evaluation (Patient-reported): Change From Baseline in Health-related Quality of Life (HR-QoL) at 12 Months (12 Visits)
Description: Patient-reported FACT-EN questionaire. Presented is the change from baseline after 12 visits/12 months. The overall total score of 43 single items was transformed to a scale from 0 to 100 (0 = worst level of well-being; 100 = highest level of well-being).
Time Frame: ICF (Baseline) up to 12 months (12 visits)
Population: FACT-En was evaluated descriptively for change from baseline of the total score using the AST population, presented for the first 12 visits. Due to death or other patients individual reasons only 4 participants were motivated to complete the FACT-En questionnaire form.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fulvestrant
Number analyzed (Participants) | 4
units on a scale | 6.0 (1.3-) [-1.3 to 13.3]

ADVERSE EVENTS:
Arm/Group | Fulvestrant
Serious Adverse Events (participants affected / at risk) | 11
Other Adverse Events (participants affected / at risk) | 32
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Fulvestrant
Tachycardia (Cardiac disorders) | 1/35
Ileus (Gastrointestinal disorders) | 2/35
Abdominal pain (Gastrointestinal disorders) | 1/35
Vomiting (Gastrointestinal disorders) | 1/35
Subileus (Gastrointestinal disorders) | 1/35
General physical health deterioration (General disorders) | 1/35
Oedema peripheral (General disorders) | 1/35
Gastroenteritis (Infections and infestations) | 1/35
Wound infection (Infections and infestations) | 1/35
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/35
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/35
Paresis (Nervous system disorders) | 1/35
Depression (Psychiatric disorders) | 1/35
Renal failure (Renal and urinary disorders) | 1/35
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1/35
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/35
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1/35
Hypertension (Vascular disorders) | 1/35
Pulmonary embolism (Vascular disorders) | 1/35
Vaginal haemorrhage (Vascular disorders) | 1/35
Deep vein thrombosis (Vascular disorders) | 1/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Fulvestrant
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/35
Abdominal pain (Gastrointestinal disorders) | 4/35
Anorexia (Metabolism and nutrition disorders) | 2/35
Ascites (Gastrointestinal disorders) | 3/35
Asthenia (General disorders) | 2/35
Back pain (Musculoskeletal and connective tissue disorders) | 2/35
Bone pain (Musculoskeletal and connective tissue disorders) | 3/35
Constipation (Gastrointestinal disorders) | 4/35
Cough (Respiratory, thoracic and mediastinal disorders) | 2/35
Diarrhoea (Gastrointestinal disorders) | 4/35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6/35
Erythema (Skin and subcutaneous tissue disorders) | 2/35
Fatigue (General disorders) | 8/35
Flatulence (Gastrointestinal disorders) | 2/35
Headache (Nervous system disorders) | 2/35
Hot flush (Vascular disorders) | 6/35
Insomnia (Psychiatric disorders) | 2/35
Lymphoedema (Vascular disorders) | 2/35
Nasopharyngitis (Infections and infestations) | 2/35
Nausea (Gastrointestinal disorders) | 9/35
Oedema peripheral (General disorders) | 3/35
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/35
Procedural site reaction (Injury, poisoning and procedural complications) | 2/35
Urinary tract infection (Infections and infestations) | 7/35
Vaginal haemorrhage (Reproductive system and breast disorders) | 4/35
Vertigo (Ear and labyrinth disorders) | 2/35
Vomiting (Gastrointestinal disorders) | 4/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No